CLINICAL TRIAL: NCT04971434
Title: Non-alcoholic Fatty Liver Response of Cardio-metabolic Risk Factors to Laser Acupuncture Versus Cupping-with-scarification
Brief Title: Fatty Liver Response of Cardio-metabolic Risk Factors to Laser Acupuncture Versus Cupping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of Physical Therapy for Cardiovascular / Respiratory Disorder and Geriatrics, Faculty of Physical Therapy, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003251
Record Dates: First submitted 2021-07-11; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Fatty Liver
MeSH Terms: conditions — Fatty Liver | interventions — Acupuncture Points

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laser (Experimental): In fatty liver patients (30 patients), a daily application of 4-minute laser (for one month, except Fridays) on acupoint number 25,40,36 of stomach meridian, acupoint number 3 of liver meridian, acupoint number 6 of spleen meridian,acupoint number 9.12,4 of conception vessel meridian, acupoint number 14 of governor vessel meridian, acupoint number 4, 11 of large intestine meridian, acupoint number 34 of gall bladder meridian
  Interventions: Device: laser stimulation for acupoints
- cupping with scarification (Experimental): In fatty liver patients (30 patients),every-two-week applied cupping (with scarification) session within one month on back of upper thorax
  Interventions: Other: cupping with scarification

INTERVENTIONS:
Device: laser stimulation for acupoints — In fatty liver patients (30 patients), a daily application of 4-minute laser (for one month, except Fridays) on acupoint number 25,40,36 of stomach meridian, acupoint number 3 of liver meridian, acupoint number 6 of spleen meridian,acupoint number 9,12,4 of conception vessel meridian, acupoint number 14 of governor vessel meridian, acupoint number 4, 11 of large intestine meridian, acupoint number 34 of gall bladder meridian
  Arms: laser
Other: cupping with scarification — In fatty liver patients (30 patients),every-two-week applied cupping (with scarification) session within one month on back of upper thorax
  Arms: cupping with scarification

SUMMARY:
Every-two-week applied cupping (with scarification) session within one month on back of upper thorax is not compared previously regarding its effect on cardio-metabolic risk factors to the daily application of laser on acupoints (for month, except Fridays) in fatty liver patients. This trial will compare the two procedure effects on cardio-metabolic risk factors in fatty liver.

DETAILED DESCRIPTION:
In fatty liver patients,every-two-week applied cupping (with scarification) session within one month on back of upper thorax for 30 patients will be compared regarding its effect on cardio-metabolic risk factors to the daily application of laser on acupoints (for month, except Fridays) of other 30 patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed Fatty liver patients by ultrasonography
* Class I obese patients

Exclusion Criteria:

* Cardiovascular and respiratory disorders/diseases.
* Autoimmune disorders/diseases.
* Pregnancy
* Other liver disorders/diseases.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — self-representation of gender identity.
Enrollment: 60 (Estimated)
Dates: Start 2021-07-11 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
high-density lipoprotein | It will be measured after 4 weeks of treatment
  serum lipid
low-density lipoprotein | It will be measured after 4 weeks of treatment
  serum lipid
cholesterol | It will be measured after 4 weeks of treatment
  serum lipid
triglyceride | It will be measured after 4 weeks of treatment
  serum lipid

SECONDARY OUTCOMES:
c reactive protein | It will be measured after 4 weeks of treatment
  it will be measured in plasma
blood glucose | It will be measured after 4 weeks of treatment
  fasting gluocse
blood pressure | It will be measured after 4 weeks of treatment
  it will be measure with manual manometer
rate of pulse | It will be measured after 4 weeks of treatment
  it will be measured at radial artery

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ismail, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Physical Therapy Cairo University, Giza, Dokki, Egypt